CLINICAL TRIAL: NCT07283185
Title: Prospective Comparison of the Carbon Footprint of Endoscopic Ultrasound (EUS) vs Magnetic Resonance Cholangiopancreatography (MRCP) for Evaluation of Suspected Choledocholithiasis
Brief Title: Prospective Comparison of the Carbon Footprint of EUS vs MRCP for Evaluation of Suspected Choledocholithiasis
Status: Recruiting | Type: Observational
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Sponsor
Other Study IDs: EUS vs MRCP-CBD1
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-10

CONDITIONS: Choledocholithiasis
MeSH Terms: conditions — Choledocholithiasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EUS: Patients scheduled for Endoscopic Ultrasound
- MRCP: Patients scheduled for Magnetic Resonance Cholangiopancreatography

SUMMARY:
MRCP and EUS are diagnostically equivalent in detecting CBD stones among patients with intermediate risk, as shown in a landmark RCT. However, MRI-based imaging is power-intensive, requiring large infrastructure and long scan durations. EUS, a less energy-consuming and portable procedure, has the added advantage of enabling same-session ERCP, reducing the need for repeat procedures.

DETAILED DESCRIPTION:
MRCP and EUS are diagnostically equivalent in detecting CBD stones among patients with intermediate risk, as shown in a landmark RCT. However, MRI-based imaging is power-intensive, requiring large infrastructure and long scan durations. EUS, a less energy-consuming and portable procedure, has the added advantage of enabling same-session ERCP, reducing the need for repeat procedures. Prior research confirms that diagnostic EUS generates significantly less CO₂e per procedure compared to radiologic imaging. This study aims to support sustainable diagnostic choices by quantifying their environmental footprint.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Intermediate likelihood of CBD stone (per ESGE)
* Undergoing either MRCP or EUS for evaluation

Exclusion Criteria:

* High or low likelihood category (per ESGE)
* Undergoing both MRCP and EUS simultaneously
* Contraindications to either modality

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (>18 years - 80years) with suspected choledocholithiasis and classified as intermediate risk per ESGE guidelines, undergoing either EUS or MRCP.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Total kg CO₂e per procedure for EUS vs MRCP. | 12 months
  Total kg CO₂e per procedure for EUS vs MRCP.

SECONDARY OUTCOMES:
Emissions | 12 months
  Emissions per accurate diagnosis Emissions broken down by source (electricity, consumables, travel) Recommendations for sustainable diagnostic practices

CONTACTS AND LOCATIONS:
Locations (1):
- AIG Hospitals, Hyderabad, Telangana, India

REFERENCES:
- [Result] • McAlister S et al. Radiology. 2021. Imaging footprint
- [Result] • Lenzen M et al. Lancet Planet Health. 2020. Health care emissions
- [Result] • Rughwani H et al. Gut. 2025. Carbon footprint of GIE
- [Result] • Jagtap N et al. Gut. 2022. EUS versus MRCP RCT